CLINICAL TRIAL: NCT01590797
Title: A Phase III, Multicenter, Randomized, Double-Blind, Placebo-Controlled Clinical Trial in China to Study the Safety and Efficacy of the Addition of Sitagliptin in Patients With Type 2 Diabetes Mellitus Who Have Inadequate Glycemic Control on Insulin Therapy, Alone or in Combination With Metformin
Brief Title: A Study in China Evaluating the Safety and Efficacy of Adding Sitagliptin to Stable Therapy With Insulin With or Without Metformin in Participants With Type 2 Diabetes Mellitus (T2DM) (MK-0431-254)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0431-254
Record Dates: First submitted 2012-05-01; First posted 2012-05-03 (Estimated); Results first posted 2015-01-27 (Estimated); Last update posted 2018-08-17 (Actual); Status verified 2018-07

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate; Insulin; Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sitagliptin (Experimental): Participants treated with sitagliptin 100 mg, once daily, for 24 weeks. All participants will be under treatment with a stable dose of insulin with or without metformin for ≥10 weeks before and throughout the study. All participants will receive placebo during the Placebo Run-in period.
  Interventions: Drug: Sitagliptin; Biological: Insulin; Drug: Metformin
- Placebo (Placebo Comparator): Participants treated with placebo matching sitagliptin, once daily, for 24 weeks. All participants will be under treatment with a stable dose of insulin with or without metformin for ≥10 weeks before and throughout the study. All participants will receive placebo during the Placebo Run-in period.
  Interventions: Drug: Placebo; Biological: Insulin; Drug: Metformin

INTERVENTIONS:
Drug: Sitagliptin — Sitagliptin 100 mg once daily for 24 weeks
  Other Names: Januvia®; MK-0431
  Arms: Sitagliptin
Drug: Placebo — Matching placebo once daily for 24 weeks
  Arms: Placebo
Biological: Insulin — Participants can be on on pre-mixed (mixture of rapid- and long-acting insulin) or intermediate- or long-acting insulin at a dose of at least 12 U/day.
Drug: Metformin — At randomization, participants will be stratified according to their use of metformin (on or not on). All participants receiving metformin will be required to be on a daily dose of metformin at least 1500 mg per day.

SUMMARY:
A study to compare safety and efficacy of sitagliptin and placebo therapy when added to stable insulin alone or in combination with metformin in participants with type 2 diabetes mellitus (T2DM). The primary hypothesis of this study is that after 24 weeks, the addition of sitagliptin compared with placebo provides greater reduction in hemoglobin A1C (HbA1C) in T2DM participants on insulin alone or in combination with metformin.

ELIGIBILITY:
Inclusion Criteria:

* has T2DM
* is currently on a stable regimen of pre-mixed, intermediate-acting, or long-acting insulin at a dose of at least 12 U/day, either alone or in combination with metformin >=1500 mg/day for ≥ 10 weeks
* has a Visit 1/Screening HbA1C between 7.5% and 11.0%
* is a male, or a female who is highly unlikely to conceive during the study and for 14 days after the last dose of study medication

Exclusion Criteria:

* has been treated with any antihyperglycemic therapies other than a protocol-required insulin (alone or with metformin) within the prior 12 weeks or has ever

been treated with a dipeptidyl peptidase-4 inhibitor or a glucagon-like peptide-1 mimetic or analogue

* is currently on treatment with daily use (one or more injections per day) of

pre-prandial short-acting or rapid-acting insulin

* has a history of 2 or more episodes of hypoglycemia resulting in seizure,

coma, or loss of consciousness, or has had recurrent episodes of hypoglycemia over the past 8 weeks

* has a history of intolerance or hypersensitivity, or has any contraindication to sitagliptin, insulin, or metformin
* is on a weight loss program and not in the maintenance phase, or has started a weight loss medication or has undergone bariatric surgery within 12 months
* has undergone a surgical procedure within 4 weeks or has planned major surgery during the study
* has a medical history of active liver disease
* has had new or worsening signs or symptoms of coronary heart disease within the past 3 months, or has acute coronary syndrome, coronary artery intervention, or stroke or transient ischemic neurological disorder
* has a diagnosis of congestive heart failure with New York Heart Association Class III - IV cardiac status
* has a systolic blood pressure ≥ 160 mmHg or a diastolic blood pressure ≥ 90 mmHg
* has human immunodeficiency virus (HIV)
* has severe peripheral vascular disease
* is currently being treated for hyperthyroidism or is on thyroid hormone therapy and has not been on a stable dose for at least 6 weeks
* has a history of malignancy ≤ 5 years before the study, except for adequately treated basal cell or squamous cell skin cancer, or in situ cervical cancer
* has a clinically important hematological disorder (such as aplastic anemia,

myeloproliferative or myelodysplastic syndromes, thrombocytopenia)

* is pregnant or breast feeding, or is expecting to conceive or donate eggs during the study, including 14 days after the last dose of study medication
* is a user of recreational or illicit drugs or has had a recent history of drug abuse

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 467 (Actual)
Dates: Start 2012-07-10 (Actual); Primary Completion 2014-06-11 (Actual); Study Completion 2014-06-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Shankar RR, Bao Y, Han P, Hu J, Ma J, Peng Y, Wu F, Xu L, Engel SS, Jia W. Sitagliptin added to stable insulin therapy with or without metformin in Chinese patients with type 2 diabetes. J Diabetes Investig. 2017 May;8(3):321-329. doi: 10.1111/jdi.12585. Epub 2016 Dec 9. PMID 27740719
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=0431-254&kw=0431-254&tab=access

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was performed with research participants at 28 study centers in China.
Groups:
- Placebo: Participants treated with placebo to sitagliptin 100 mg, once daily, for 24 weeks. All participants will be under treatment with a stable dose of insulin with or without metformin for ≥10 weeks before and throughout the study. All participants will receive placebo during the Placebo Run-in period.
Period: Overall Study
Arm/Group | Sitagliptin | Placebo
Started | 234 | 233
Completed | 217 | 217
Not Completed | 17 | 16
Not completed — Adverse Event | 4 | 3
Not completed — Lack of Efficacy | 0 | 2
Not completed — Lost to Follow-up | 0 | 1
Not completed — Protocol Violation | 4 | 1
Not completed — Withdrawal by Subject | 7 | 5
Not completed — Other Protocol Specified Criteria | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sitagliptin | Placebo | Total
Number analyzed (Participants) | 234 | 233 | 467
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.6 (8.4) | 56.7 (9.1) | 57.6 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 104 | 117 | 221
  Male | 130 | 116 | 246

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hemoglobin A1C (HbA1C) Levels at Week 24 in Participants Receiving Insulin Alone or in Combination With Metformin
Time Frame: Baseline and Week 24
Population: The Full Analysis Set (FAS) consisted of all randomized participants receiving insulin alone or in combination with metformin, took at least one dose of study treatment, had at least one observation for the analysis endpoint subsequent to the first dose of study treatment, and had baseline data for the analysis endpoint.
Measure: Least Squares Mean (95% Confidence Interval); unit: A1C %
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 223 | 219
A1C % | -0.67 [-0.79 to -0.55] | -0.32 [-0.44 to -0.20]
Statistical Analysis 1: Comparison: Sitagliptin vs Placebo; Test type: Superiority or Other; p < 0.001, Robust Regression; Robust regression using M-estimation with terms for treatment and the metformin stratum and type of insulin, and baseline A1C (%) as a covariate; Mean Difference (Final Values) = -0.34, 95% CI 2-sided [-0.50 to -0.19]

2. Secondary Outcome: Change From Baseline in HbA1C Levels at Week 24 in Participants Receiving Insulin in Combination With Metformin
Time Frame: Baseline and Week 24
Population: The FAS consisted of all randomized participants receiving insulin in combination with metformin, took at least one dose of study treatment, had at least one observation for the analysis endpoint subsequent to the first dose of study treatment, and had baseline data for the analysis endpoint.
Measure: Least Squares Mean (95% Confidence Interval); unit: A1C %
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 109 | 104
A1C % | -0.72 [-0.89 to -0.55] | -0.34 [-0.51 to -0.17]
Statistical Analysis 1: Comparison: Sitagliptin vs Placebo; Test type: Superiority or Other; p = 0.002, Robust Regression; Robust regression using M-estimation with terms for treatment and type of insulin, and baseline A1C (%) as a covariate; Mean Difference (Final Values) = -0.38, 95% CI 2-sided [-0.61 to -0.14]

3. Secondary Outcome: Change From Baseline in 2-Hour Post Meal Glucose Levels at Week 24 in Participants Receiving Insulin Alone or in Combination With Metformin
Time Frame: Baseline and Week 24
Population: The FAS consisted of all randomized participants receiving insulin alone or in combination with metformin, took at least one dose of study treatment, had at least one observation for the analysis endpoint subsequent to the first dose of study treatment, and had baseline data for the analysis endpoint.
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 209 | 203
mg/dL | -47.9 [-57.0 to -38.8] | -21.3 [-30.3 to -12.3]
Statistical Analysis 1: Comparison: Sitagliptin vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; ANCOVA model with terms for treatment and the metformin stratum and type of insulin, and baseline 2-hr Post- Meal Glucose (mg/dL) as a covariate; Mean Difference (Final Values) = -26.5, 95% CI 2-sided [-38.4 to -14.7]

4. Primary Outcome: Number of Participants With One or More Adverse Events
Description: An adverse event (AE) is defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it is considered related to the medical treatment or procedure, that occurs during the course of the study.
Time Frame: Up to Week 26
Population: The All Patients as Treated (APaT) population consisted of all randomized participants who received at least one dose of study treatment. Participants were included in the treatment group corresponding to the study treatment they actually received for the analysis of safety data.
Measure: Number; unit: Participants
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 234 | 233
Participants | 126 | 116

5. Primary Outcome: Number of Participants Discontinuing Study Medication Due to an AE
Description: An AE is defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it is considered related to the medical treatment or procedure, that occurs during the course of the study.
Time Frame: Up to Week 24
Population: The APaT population consisted of all randomized participants who received at least one dose of study treatment. Participants were included in the treatment group corresponding to the study treatment they actually received for the analysis of safety data.
Measure: Number; unit: Participants
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 234 | 233
Participants | 4 | 2

ADVERSE EVENTS:
Time Frame: Up to Week 26
Description: The APaT population consisted of all randomized patients who received at least one dose of study treatment. Participants were included in the treatment group corresponding to the study treatment they actually received for the analysis of safety data.
Arm/Group | Sitagliptin | Placebo
Serious Adverse Events (participants affected / at risk) | 4/234 | 9/233
Other Adverse Events (participants affected / at risk) | 83/234 | 68/233
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sitagliptin (N=234) | Placebo (N=233)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric polyps (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diabetic foot infection (Infections and infestations) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 1 (1)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Vertebrobasilar insufficiency (Nervous system disorders) | 0 (0) | 1 (1)
Diabetic nephropathy (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure chronic (Renal and urinary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sitagliptin (N=234) | Placebo (N=233)
Blood glucose increased (Investigations) | 16 (40) | 13 (32)
Upper respiratory tract infection (Infections and infestations) | 12 (13) | 11 (13)
Hypoglycaemia (Metabolism and nutrition disorders) | 65 (173) | 52 (150)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the sponsor as confidential must be deleted prior to submission.